CLINICAL TRIAL: NCT05402670
Title: Gastric Mucosal Changes in Patients With Dermatomyositis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0656
Record Dates: First submitted 2021-11-08; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Gastric Mucosal Manifestations in Patients With Dermatomyositis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dermatomyositis group: patient with dermatomyositis
- control group: health check-up population

INTERVENTIONS:
Other:

SUMMARY:
There are a large number of reports in the literature that patients with dermatomyositis often have various malignant tumors, and reports of gastric cancer are not rare. At present, the widely recognized gastric cancer occurrence patterns are: normal gastric mucosa-chronic superficial gastritis-chronic atrophic gastritis-intestinal metaplasia-dysplasia-gastric cancer, so the research about the gastric mucosal performance of patients with dermatomyositis is clinically meaningful

ELIGIBILITY:
Inclusion Criteria:

* 1、18-70years old，no gender limit. 2、Clinical diagnosis of dermatomyositis. 3、dermatomyositis group conform to 1 and 2，control group conform to 1 .

Exclusion Criteria:

* Contraindications for gastroscopy.

  * Past history of malignant tumors of the esophagus and stomach and or history of surgery.

    * Pregnant or lactating women. ④ Participated in other clinical studies within 3 months. ⑤Patients cannot express their main complaints correctly and cannot cooperate with the research.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dermatomyositis patients in the Department of Rheumatology, the Second Affiliated Hospital of Zhejiang University School of Medicine。 Healthy people undergoing physical examination at the Physical Examination Center of the Second Affiliated Hospital of Zhejiang University School of Medicine。
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Gastric mucosal manifestations | 1 year
  Normal gastric mucosa、chronic superficial gastritis、chronic atrophic gastritis、intestinal metaplasia、dysplasia、gastric cancer、gastric ulcer and so on

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No